CLINICAL TRIAL: NCT01289522
Title: Phase II Study of Cetuximab, Docetaxel and Cisplatin as First-line Treatment in Patients With Metastatic or Recurrent Head and Neck Squamous Cell Carcinomas - GORTEC 2008-03 TPEx
Brief Title: Chemotherapy With Cetuximab in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Acronym: TPEx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2008-03 TPEx; 2008-004869-25 (EudraCT Number)
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2016-10

CONDITIONS: Squamous Cell Head and Neck Carcinoma; Recurrent or Metastatic Disease
Keywords: Squamous cell carcinoma of the head and neck; recurrent or metastatic; first line chemotherapy; cetuximab; docetaxel; cisplatin; antineoplastic agents; First Line Palliative Treatment
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Recurrence; Neoplasm Metastasis | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cetuximab (Experimental): Patients receive four cycles of chemotherapy comprising cetuximab IV plus docetaxel IV over 1 hour and cisplatin IV over 2 hours on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. After completion of the fourth cycle of chemotherapy, patients receive a maintenance therapy with cetuximab every 2 weeks. Treatment will be continued until disease progression or unacceptable toxicities according
  Interventions: Biological: cetuximab IV; Other: Biopsies

INTERVENTIONS:
Biological: cetuximab IV — * Cetuximab 400 mg/m² over 120 minutes on day 1 of cycle 1 only.
  * Cetuximab dose will be 250 mg/m² IV over 60 minutes weekly on subsequent administrations during the four cycles of chemotherapy.
  * Cetuximab dose will be 500mg/m2 IV every 2 weeks during the maintenance therapy.
  Drug: Cisplatin IV : 75 mg/m2 intravenous every 3 weeks for 4 cycles
  Drug: Docetaxel IV : 75 mg/m2 intravenous every 3 weeks for 4 cycles
  G-CSF support with lenograstim 150 microg./m2/day is delivered after each cycle of chemotherapy.
Other: Biopsies — No intervention, only biopsy for translational project.

SUMMARY:
PURPOSE: Cetuximab with platinum and 5FU is now the standard combination as first-line treatment in patients with metastatic or recurrent Head and Neck squamous cell carcinomas. Cetuximab and taxane combinations have demonstrated promising activity in Head and Neck cancer. This phase II trial is studying new cetuximab, docetaxel and cisplatin combination named TPEx as first-line treatment in this setting.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy of TPEx combination in patients with head and neck cancer in term of objective response rate (RECIST, see statistical consideration) Secondary
* To assess toxicities of TPEx combination
* Determine the efficacy of TPEx combination in patients with head and neck cancer: Best Overall Response , progression-free survival and survival.
* Translational research objective:To better understand the mechanisms of chemoresistance and to identify biomarkers by the analysis of the tumor biopsies (RNA, gene expression profile) and protein profile (plasma samples). Exploratory analyses.

OUTLINE: This is an open-label phase II, multicenter study. Patients receive four cycles of chemotherapy comprising cetuximab IV plus docetaxel IV over 1 hour and cisplatin IV over 2 hours on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. After completion of the fourth cycle of chemotherapy, patients receive a maintenance therapy with cetuximab every 2 weeks. Treatment will be continued until disease progression or unacceptable toxicities according to the patient or the investigator. Tumor check-up will be performed every 6 weeks. This study will allow translational research with blood sample and biopsies at baseline before any treatment, during the treatment with TPEx combination (week 6).,After completion of study treatment, patients are followed every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the oral cavity, larynx, oropharynx or hypopharynx
* Recurrent disease, incurable disease as determined by surgery or radiation, or metastatic disease
* Measurable or evaluable disease
* Age > 18 years and <= 70 years
* WHO performance status 0 or 1
* Absolute neutrophil count > 1,500/mm3
* Platelets > 150,000/mm3
* Total Bilirubin <= institutional upper limit of normal
* Aspartate aminotransferase < 1.5 X institutional upper limit of normal
* Alanine aminotransferase < 1.5 X institutional upper limit of normal
* Alkaline phosphatase < 2.5 X institutional upper limit of normal
* creatinine clearance > 60 mL/min
* Signed informed consent
* Women of child-bearing potential and men must be willing and able practice adequate contraception prior to study entry and for the duration of study treatment

Exclusion Criteria:

* Previous chemotherapy. Chemotherapy given as part of initial curative therapy and completed more than 6 months before inclusion is allowed
* Previous treatment with total doses of cisplatin > 300 mg/ m2
* Patients must not have any co-existing disease that would preclude cisplatin administration, such as peripheral neuropathy or renal failure
* Surgery (excluding biopsy) or radiotherapy within 4 weeks prior to study entry
* Nasopharyngeal carcinoma, or cancer of sinusal cavities
* Active infection including tuberculosis or HIV positive patient
* Other malignancy within last 5 years except for non-melanoma skin cancer
* No other investigational agent within 30 days prior to study entry
* No other concurrent chemotherapy, immunotherapy, antitumor hormonal therapy (excluding contraceptives and replacement steroids), radiotherapy, or experimental medications
* No prior anti EGFR therapy
* No known brain metastases
* Uncontrolled intercurrent illness that would prevent delivery of protocol therapy
* Patients with a prior history of basal cell carcinoma of the skin or in situ carcinoma of the cervix must have been curatively treated and must have remained disease free for 5 years post diagnosis
* No history of hypersensitivity reaction to drugs on study
* No unstable angina or myocardial infarction within the past 12 months
* No symptomatic congestive heart failure or New York Heart Association (NYHA) class II-IV heart disease
* No serious uncontrolled cardiac arrhythmia
* No other prior or concomitant squamous cell carcinoma
* No other prior or concomitant cancer, except curatively treated basal carcinoma of the skin or in situ cervical cancer, for which the patient has been curatively treated and remains disease-free for the past 5 years
* Patient is pregnant or lactating
* Patients must not have any co-existing condition that would preclude full compliance with the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel GUIGAY, Study Chair — GORTEC
Locations (14):
- Belgium (3):
  - Cliniques Universitaires, Brussels
  - Clinique Sainte Elisabeth, Namur
  - Clinique universitaire de Mont Godinne UCL, Yvoir
- France (11):
  - Hôpital Saint André, Bordeaux
  - Centre Jean Perrin,, Clermont-Ferrand
  - Centre G-F Leclerc, Dijon
  - Centre Hospitalier de la Dracénie, Draguignan
  - Centre Hospitalier de Bretagne Sud, Lorient
  - Centre Léon Bérard, Lyon
  - Hôpital de la Timone, Marseille
  - Centre Henri Becquerel, Rouen
  - Hôpital Foch, Suresnes
  - CHU Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Guigay J, Fayette J, Dillies AF, Sire C, Kerger JN, Tennevet I, Machiels JP, Zanetta S, Pointreau Y, Bozec Le Moal L, Henry S, Schilf A, Bourhis J. Cetuximab, docetaxel, and cisplatin as first-line treatment in patients with recurrent or metastatic head and neck squamous cell carcinoma: a multicenter, phase II GORTEC study. Ann Oncol. 2015 Sep;26(9):1941-1947. doi: 10.1093/annonc/mdv268. Epub 2015 Jun 24. PMID 26109631

RESULTS

PARTICIPANT FLOW:
Groups:
- Cetuximab: cetuximab IV: - 400 mg/m² over 120 minutes on day 1 of cycle 1 only.
  * 250 mg/m² over 60 minutes weekly on subsequent administrations
  * 500mg/m2 every 2 weeks during the maintenance therapy. Drug: -Cisplatin IV : 75 mg/m2 every 3 weeks for 4 cycles
  * Docetaxel IV : 75 mg/m2 every 3 weeks for 4 cycles G-CSF support mandatory after each cycle of chemotherapy. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. After completion of the 4th cycle of chemotherapy, patients receive a maintenance therapy with cetuximab every 2 weeks.
Period: Overall Study
Arm/Group | Cetuximab
Started | 54
Completed | 43
Not Completed | 11

BASELINE CHARACTERISTICS:
Groups:
- Cetuximab: Patients receive four cycles of chemotherapy comprising cetuximab IV plus docetaxel IV over 1 hour and cisplatin IV over 2 hours on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. After completion of the fourth cycle of chemotherapy, patients receive a maintenance therapy with cetuximab every 2 weeks. Treatment will be continued until disease progression or unacceptable toxicities according cetuximab IV: - 400 mg/m² over 120 minutes on day 1 of cycle 1 only.
  * 250 mg/m² IV over 60 minutes weekly on subsequent administrations during the four cycles of chemotherapy.
  * 500mg/m2 IV every 2 weeks during the maintenance therapy.
  Drug: Cisplatin IV : 75 mg/m2 every 3 weeks for 4 cycles Drug: Docetaxel IV : 75 mg/m2 every 3 weeks for 4 cycles
  G-CSF support with lenograstim 150 microg./m2/day is delivered after each cycle of chemotherapy.
  Biopsies: No intervention, only biopsy for translational project.
Arm/Group | Cetuximab
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 52
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 57.8 [28.9 to 69.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 52
Region of Enrollment [Number; unit: participants]
  Belgium | 8
  France | 46

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response Rate
Description: The objective tumor response rate is evaluated every 6 weeks according to RECIST criteria.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT-scan or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: 12 weeks (after completion of the 4th cycle of chemotherapy)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cetuximab: Patients receive four cycles of chemotherapy comprising cetuximab IV plus docetaxel IV over 1 hour and cisplatin IV over 2 hours on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. After completion of the fourth cycle of chemotherapy, patients receive a maintenance therapy with cetuximab every 2 weeks. Treatment will be continued until disease progression or unacceptable toxicities according
  cetuximab IV: - 400 mg/m² over 120 minutes on day 1 of cycle 1 only.
  * 250 mg/m² IV over 60 minutes weekly on subsequent administrations during the four cycles of chemotherapy.
  * 500mg/m² IV every 2 weeks during the maintenance therapy. Drug: Cisplatin IV : 75 mg/m² every 3 weeks for 4 cycles Drug: Docetaxel IV : 75 mg/m² every 3 weeks for 4 cycles
  G-CSF support with lenograstim 150 microg/m²/day is delivered after each cycle of chemotherapy.
  Biopsies: No intervention, only biopsy for translational project.
Arm/Group | Cetuximab
Number analyzed (Participants) | 54
percentage of participants | 44 [30.9 to 58.6]

2. Secondary Outcome: Grade 1 to 5 Toxicity
Description: All grade 1 to 5 toxicity are registered during treatment. Patients have weekly clinical and biological examination.
Time Frame: 24 weeks (average)
Measure: Number; unit: percentage of events
Arm/Group | Cetuximab
Number analyzed (Participants) | 54
percentage of events | 50

3. Secondary Outcome: Best Overall Response
Description: Tumor response is evaluated every 6 weeks according to RECIST criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions, Stable Disease (SD); Best overall Response = CR + PR + SD.
Time Frame: 12 weeks
Population: 2 patients not assessable for response at 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of Best overall ORR
Arm/Group | Cetuximab
Number analyzed (Participants) | 52
percentage of Best overall ORR | 53.7 [39.6 to 67.4]

4. Secondary Outcome: Progression-free Survival
Time Frame: 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival
Time Frame: 1 year
Reporting Status: Not Posted

6. Secondary Outcome: Biomarkers
Time Frame: two years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Cetuximab
Serious Adverse Events (participants affected / at risk) | 15/54
Other Adverse Events (participants affected / at risk) | 35/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab (N=54)
arterial rupture (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Oral intake reduced (Metabolism and nutrition disorders) | 1 (1)
Acute alcoholic hepatitis (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Central line infection (Infections and infestations) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1)
haemoptysis (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab (N=54)
anemia (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Hyponatremia (Investigations) | 1 (1)
hypokalemia (Investigations) | 2 (2)
diarrhea (Gastrointestinal disorders) | 2 (2)
oral mucositis (Gastrointestinal disorders) | 3 (3)
fever (General disorders) | 1 (1)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
renal failure (Renal and urinary disorders) | 1 (1)
hearing loss (Ear and labyrinth disorders) | 1 (1)
skin toxicities (Skin and subcutaneous tissue disorders) | 7 (7)
neutropenia (Blood and lymphatic system disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less